CLINICAL TRIAL: NCT04416308
Title: COVID 19 : Seroprevalence Study of Anti SRAS-CoV-2 Antibodies in GHT Employees in Haute Bretagne
Brief Title: COVID 19 : Seroprevalence Study of Anti SRAS-CoV-2 Antibodies in GHT Employees in Haute Bretagne (AntiCoV-HB)
Acronym: AntiCoV-HB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Collaborators: Fonds NOMINOE (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 35RC20_9716
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Coronavirus
Keywords: Covid 19, SRAS-CoV-2
MeSH Terms: conditions — Coronavirus Infections; COVID-19 | interventions — Hematologic Tests

STUDY DESIGN:
Intervention Model Description: This is a multi-center cross-sectional survey at risk and minimal constraints, among GHT Haute Bretagne employees in order to know the prevalence of the presence of anti-SARS-CoV-2 antibodies.
  For a sample of employees with no additional prospective follow-up will be done on D30 and D90.
Who Masked: Outcomes Assessor
Masking Description: For the first 30 employees a second test will be carried out a few minutes after the first test by another nurse blinded to the result of the first test in order to estimate the agreement between - observers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Seroprevalence survey (Other): NG Test + short self-questionnaire (except validation survey and detailed survey)
  Interventions: Diagnostic Test: NG test; Behavioral: Self-questionnary
- Validation test of the NG test survey (Other): Blood test + NG test + detailed self-questionnaire
  Interventions: Diagnostic Test: NG test; Diagnostic Test: Blood test; Behavioral: Self-questionnary
- Detailed Survey (Other): NG test + self-questionnaire complementary to the short questionnaire
  Interventions: Diagnostic Test: NG test; Behavioral: Self-questionnary
- Prevalence monitoring (2 population samples) (Other): Participants having presented a certain or probable COVID: acts of the validation test survey, + follow-up questionnaire,+ blood test + NG test, on D30 and D90
  Others Participants : drawn by lot: acts of the seroprevalence survey, + follow-up questionnaire + NG test, on D90
  Interventions: Diagnostic Test: NG test; Diagnostic Test: Blood test; Behavioral: Self-questionnary

INTERVENTIONS:
Diagnostic Test: NG test — rapid diagnosis Covid 19
Diagnostic Test: Blood test — sample
  Arms: Prevalence monitoring (2 population samples); Validation test of the NG test survey
Behavioral: Self-questionnary — behavioral survey

SUMMARY:
Since the start of this epidemic, numerous clinical and fundamental studies have been conducted to best adapt the individual management of COVID-19 cases [1-6]. In parallel with this work, it is necessary to better understand the characteristics of the epidemic in the general population but also in the population working in healthcare settings more exposed to SARS-CoV-2. Seroprevalence studies are therefore particularly useful in order to understand the collective immunization rate and the factors that can explain this immunization.

DETAILED DESCRIPTION:
The first cases of the new coronavirus disease 2019 (COVID-19) due to the SARS-CoV-2 virus were reported in December 2019 in Wuhan, China. Since that date, a significant circulation of the virus around the world has been observed, justifying that WHO described the situation as pandemic on March 11.

Since the start of this epidemic, numerous clinical and fundamental studies have been conducted to best adapt the individual management of COVID-19 cases. In parallel with this work, it is necessary to better understand the characteristics of the epidemic in the general population but also in the population working in healthcare settings more exposed to SARS-CoV-2. Seroprevalence studies are therefore particularly useful in order to understand the collective immunization rate and the factors that can explain this immunization. In the general population, only one recent study in France, in the Oise, one of the first clusters in France, reports a seroconversion rate of 35% in the area concerned [7]. This study used three different tests (ELISA, S-FLOW, LIPS assays) to define seroconversion (people were considered positive if at least one of the tests reported the presence of Anti SARS CoV 2 Antibodies).

The proportion of people infected in Brittany, estimated by modeling work, would be 1.8% [1.1% -3.3%]. At the present time, no data exist to our knowledge on the seroprevalence of anti SARS-CoV-2 antibodies in healthcare populations. Many serological tests are currently being validated. The Rennes University Hospital, thanks to the support of the NOMINOE fund, will offer all employees of the territory hospital group (GHT) Haute-Bretagne to participate in this seroprevalence study using the serological test from the company NG-Biotech. It is a device of the type "rapid serological diagnostic orientation test (TROD)" which can be carried out outside medical biology laboratories by a doctor / pharmacist who is not a biologist or a nurse. This test provides a result in about fifteen minutes. The NG-Biotech test has a CE / IVD mark (pending opinion from the Institut Pasteur). An assessment of the sensitivity and specificity of the test was carried out at the CHU Kremlin Bicêtre and CHU Paul Brousse. From a sample of 101 COVID-19 patients (diagnosed by RT-PCR on nasopharyngeal or pulmonary samples) and 50 negative controls (30 pre-pandemic sera from September and October 2017 and 20 sera from patients tested COVID- 19 negative by RT-PCR without any symptoms for more than 15 days) a sensitivity of 97% [88.7% - 99.4%] and a specificity of 100% [91.1% -100%] were obtained 15 days after the first signs of COVID-19 patients. If the validity of the test is very good in this study, its main limitation is that it was carried out with a group of COVID-19 patients who were in the vast majority hospitalized (84% of patients) and therefore not representative of pauci or asymptomatic patients .

Consequently, given the absence of consolidated data on the immune response based on clinical pictures, it is relevant to continue validation in a population of employees in which we wish to carry out this seroprevalence study and where the majority of infections did not lead to hospitalization. In addition, it is also necessary to obtain other data, in particular concerning the inter-observer reproducibility of the test which has not yet been studied. The need to validate the test in pauci or asymptomatic populations and to obtain reproducibility data was underlined in the opinion of the HAS on the methods for evaluating the performance of serological tests detecting antibodies directed against SARS-CoV -2.

ELIGIBILITY:
Inclusion Criteria:

* Employees of voluntary establishments of GHT Haute-Bretagne
* Employees over the age of 18
* Having signed a free, informed and written consent.

Exclusion Criteria:

* Employees subject to legal protection (safeguard of justice, guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9453 (Actual)
Dates: Start 2020-05-29 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-10-12 (Actual)

PRIMARY OUTCOMES:
rate of presence of anti-SARS-CoV-2 antibodies (Ig G _ Ig M) among employees working in a GHT Haute Bretagne health establishment. | at inclusion visit
  Rate of presence

SECONDARY OUTCOMES:
a) Validation of the Biotech NG test: | at inclusion visit
  Sensitivity
a) Validation of the Biotech NG test: | at inclusion visit
  Specificity
a) Validation of the Biotech NG test: Agreement between observers (kappa coefficient) for IgG | at inclusion visit
  agreement between observers (kappa coefficient)
a) Validation of the Biotech NG test: Agreement between observers (kappa coefficient) for IgM. | at inclusion visit
  agreement between observers (kappa coefficient)
b) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  Demographic characteristics (age, sex)
b) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  - Professional characteristics (establishment, profession, service).
b) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  - Management of confirmed or probable COVID-19 patients
b) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  - From contact with confirmed or probable COVID-19 professionals.
b) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  - From contact in his personal circle with COVID-19 confirmed or probable persons.
b) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  - Episodes of symptoms suggestive of COVID-19
b) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  - The existence of a chronic immunomodulatory pathology
b) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  - The existence of smoking
c) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  - The use of materials adapted to good hygiene practices
c) Risk of presence of anti SARS-CoV-2 antibodies in function: | At inclusion visit
  - Service organization
d) Description of the experience and behavioral changes related to the epidemic, | at Day 0
  depending on the work sector (COVID dedicated or not) and depending on the profession:
  - Rate of employees who changed their tobacco consumption
d) Description of the experience and behavioral changes related to the epidemic, | at Day 0
  depending on the work sector (COVID dedicated or not) and depending on the profession:
  - Description of the reasons for modifying tobacco consumption
d) Description of the experience and behavioral changes related to the epidemic, | at Day 0
  depending on the work sector (COVID dedicated or not) and depending on the profession:
  - Rate of employees who changed their alcohol consumption
d) Description of the experience and behavioral changes related to the epidemic, | at Day 0
  depending on the work sector (COVID dedicated or not) and depending on the profession:
  - Description of the reasons for modification of alcohol consumption
d) Description of the experience and behavioral changes related to the epidemic, | at Day 0
  depending on the work sector (COVID dedicated or not) and depending on the profession:
  - Rate of employees who have changed their eating habits
d) Description of the experience and behavioral changes related to the epidemic, | at Day 0
  depending on the work sector (COVID dedicated or not) and depending on the profession:
  - Description of sleep changes
d) Description of the experience and behavioral changes related to the epidemic, | at Day 0
  depending on the work sector (COVID dedicated or not) and depending on the profession:
  - Description of lived experience and perceived stress
e) Evolution of seroprevalence over time: | At Day30
  For employees identified as COVID "certain or probable"
  * Percentage of employees with antibodies (IgG and IgM) against SARS CoV-2 on D30 and D90.
e) Evolution of seroprevalence over time: | At Day 90
  For employees identified as COVID "certain or probable"
  * Evolution of the kinetics of antibodies (IgG and IgM) against SARS CoV-2 on D30 and D90.
e) Evolution of seroprevalence over time: | At Day 90
  For the random sample of employees with follow-up on D90: Percentage of employees with antibodies (IgG and IgM) against SARS CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Christophe PARIS, MD, Principal Investigator — CHU Rennes
Locations (9):
- France (9):
  - CENTRE HOSPITALIER de VITRE_ Saint Jean (La Guerche), La Guerche-de-Bretagne, La Guerche-de-Bretagne
  - Centre Hospitalier de Fougeres, Fougères
  - Centre Hospitalier Grand Fougeray, Grand-Fougeray
  - Centre Hospitalier de La Roche Aux Fees, Janzé
  - Centre Hospitalier Montfort-Sur-Meu, Montfort-sur-Meu
  - Centre Hospitalier de Redon Carentoir, Redon
  - Chu Rennes, Rennes
  - Centre Hospitalier St Meen Le Grand, Saint-Méen-le-Grand
  - CENTRE HOSPITALIER VITRE_Simone Veil, Vitré

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Garlantezec R, Heslan C, Tadie E, Tattevin P, Thibault V, Paris C. A lateral flow immunoassay test performance in SARS-CoV-2 seroprevalence surveys: a validation study among healthcare workers. Emerg Microbes Infect. 2020 Dec;9(1):2547-2549. doi: 10.1080/22221751.2020.1852893. PMID 33206004
- [Result] Garlantezec R, Tadie E, Heslan C, Gary-Bobo P, Oumari S, Saade A, Sitruk A, Tattevin P, Thibault V, Paris C; AntiCOV-HB* working group. SARS-CoV-2 seroprevalence and antibodies persistence among health care workers after the first COVID-19 wave in nine hospitals in Western France. Infect Dis Now. 2022 Nov;52(8):447-452. doi: 10.1016/j.idnow.2022.09.004. Epub 2022 Sep 13. PMID 36108975
- [Result] Paris C, Tadie E, Heslan C, Gary-Bobo P, Oumari S, Saade A, Sitruk A, Wild P, Thibault V, Tattevin P, Garlantezec R. Risk factors for SARS-CoV-2 infection among health care workers. Am J Infect Control. 2022 Apr;50(4):375-382. doi: 10.1016/j.ajic.2021.11.001. Epub 2021 Nov 12. PMID 34774895